CLINICAL TRIAL: NCT00178789
Title: Prospective Observational Trial of Point-of-Care, Limited Ultrasonography (PLUS) for Lower Extremity Deep Venous Thrombosis in the Emergency Department: The Sonography Outcomes Assessment Program (SOAP-4 Trial)
Brief Title: Sonography Outcomes Assessment Program for Lower Extremity Deep Venous Thrombosis
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Other Study IDs: HSC-MS-05-0011
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2007-05-23 (Estimated); Status verified 2007-05

CONDITIONS: Deep Venous Thrombosis
Keywords: Deep Venous Thrombosis; Blood Clot; Lower Extremity; Sonography
MeSH Terms: conditions — Venous Thrombosis; Thrombosis

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Currently, most emergency physicians have limited access to obtaining formal radiology ultrasound studies, particularly overnight. Many are forced to adopt risky and expensive strategies in managing their patients with suspected deep venous thrombosis (DVT) who present during off-hours: for low risk patients, discharging without anticoagulation and arranging for outpatient studies; for moderate to high risk patients, empirically anticoagulating and admitting to the hospital to await definitive testing. If emergency physicians could reliably perform an accurate ultrasound exam for DVT, such risks could be obviated.

This is a prospective, observational cohort study assessing the accuracy of emergency physician diagnosis of proximal DVT using compact ultrasound equipment and a simplified compression technique. The value of color flow doppler and augmentation will also be assessed. Outcomes (sensitivity, specificity, positive likelihood ratio and negative likelihood ratio) will be assessed at 30 days.

Prior to enrolling patients in the study, emergency physicians will undertake a 2 hour training course on the performance of the simplified compression technique for the diagnosis of lower extremity DVT. Emergency physicians will perform the DVT ultrasound exam on study subjects with suspected DVT. Clinical management of the study subjects will not be altered; all subjects will proceed to receive a formal DVT ultrasound study by the radiology department which will serve as the criterion reference for the study.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

  1. Presenting signs and symptoms sufficiently suspicious for lower extremity DVT to warrant a formal radiology study in the opinion of the treating physician AND EITHER 2a. Moderate or high pre-test clinical probability of DVT (Wells Criteria) OR 2b. Low pre-test clinical probability of DVT with a positive D-dimer

Exclusion Criteria:

* Exclusion criteria:

  1. Documented lower extremity DVT within the past 60 days
  2. Anatomic abnormality that, in the judgment of the investigator, would preclude imaging of both femoral and popliteal veins on the affected leg (i.e. above-knee amputation or severe scarring from intravenous drug abuse in the inguinal area)
  3. Patient below the age of 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2005-09; Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory M Press, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann Hospital Emergency Department, Houston, Texas, United States